CLINICAL TRIAL: NCT02442544
Title: Effect of Prebiotic Fiber on Gut Microbiota, Intestinal Permeability and Glycemic Control in Children With Type 1 Diabetes: A Pilot Randomized, Double Blind, Placebo Controlled Study
Brief Title: Prebiotic Fiber Supplement in T1DM Children
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Carol Huang, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OFSDM1
Record Dates: First submitted 2015-03-10; First posted 2015-05-13 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): maltodextrin 3.3 g orally/ day for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Prebiotic (Experimental): 1:1 oligofructose: inulin 8 g orally /day for 12 weeks
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — 1:1 oligofructose: inulin 8 g orally /day
  Other Names: OFS
  Arms: Prebiotic
Dietary Supplement: Placebo — maltodextrin 3.3g orally/day
  Arms: Placebo

SUMMARY:
The gut microbiome is increasingly recognized as a contributor to disease states. In type 1 diabetes, alterations in gut microbiota may be linked to changes in intestinal permeability, inflammation and insulin resistance. Prebiotic fiber is a dietary supplement that alters gut microbiota and could potentially improve insulin sensitivity in children with type 1 diabetes. This pilot study aims to determine the feasibility of a 12-week dietary intervention with prebiotic fiber in children with type 1 diabetes. The investigators hypothesize that consumption of prebiotic fiber will alter gut microbiota and intestinal permeability, leading to improved glycemic control. Prebiotic fiber is a potentially novel, inexpensive, low-risk treatment addition for type 1 diabetes that may improve glycemic control by changes in gut microbiota, gut permeability and inflammation.

DETAILED DESCRIPTION:
At baseline, each subject will complete a demographic questionnaire (age, gender, date of type 1 diabetes diagnosis, current medications, other medical conditions, number of episodes of severe hypoglycemia and diabetic ketoacidosis since diagnosis of type 1 diabetes) and an anthropometric data form (height, weight, body mass index). A baseline stool sample will be collected at home. One tablespoon of stool will be placed in a pre-labelled sterile conical tube, placed in a biohazard bag and stored in the home freezer (-20°C). Stool samples will be brought to the laboratory on ice within 3 days from collection and stored at -80°C until analysis. Subjects will have a baseline blood sample drawn for HbA1c, C-peptide, and inflammatory markers (IL-6, IFN-γ, TNF-α, and IL-10), GLP1 and GLP2. An intestinal permeability test will be performed as described below.

Subjects will be randomized to receive either placebo (maltodextrin 3.3 g orally/ day) or prebiotic fiber (1:1 oligofructose: inulin 8 g orally /day). Both are approved as food ingredients in Canada and not regulated as natural health products. Dr. Reimer has a 'no objection' letter from Health Canada and has previously used these in a clinical trial (14).

Both prebiotic fiber and placebo come in a powder form in a pre-measured packet. Subjects will be instructed to mix the packet with 250 mL water until dissolved and to take 15-20 minutes prior to their evening meal. For the first two weeks, subjects will be asked to only take half of the dose in order to minimize GI side effects and then they will take the full dose for the remaining 10 weeks. Subjects will be asked to record any diabetes related adverse reactions (ie. severe hypoglycemia and diabetic ketoacidosis). At the end of the 12 weeks (3months), subjects will be asked to submit a second stool sample and repeat baseline blood tests and intestinal permeability testing. Subjects will be asked to return any remaining packets of placebo or prebiotic in order to assess for compliance. A third stool sample, intestinal permeability testing and blood sample (HbA1c, C-peptide, inflammatory markers (IL-6, IFN-γ, TNF-α, and IL-10), GLP1 and GLP2) will be done at 6 months follow up. Telephone contact from a member of the research team (research assistant or PI) will occur monthly to encourage compliance and recording of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 - 17 years old
2. Diagnosed with type 1 diabetes for at least one year
3. HbA1c <10% for 6 month prior to start of trial

Exclusion Criteria:

1. Subjects with another chronic medical condition that could affect gut microbiota (examples: Crohn's disease, cystic fibrosis, irritable bowel syndrome, etc.)
2. Subjects taking medications or supplements that could affect gut microbiota (examples: antibiotics, probiotics, prebiotics, laxatives, etc.)
3. Subjects with a positive celiac disease screen

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (serum hemoglobin A1c) | 3 month after start of trial
  measure serum level of hemoglobin A1c

SECONDARY OUTCOMES:
Gut microbiota composition (mRNA in stool) | 3 month after start of trial
  measure mRNA in stool
Gut microbiota composition (mRNA in stool) | 6 month after start of trial
  measure mRNA in stool
Glycemic control (as measured by serum hemoglobin A1c) | 6 month after start of trial
  measure serum level of hemoglobin A1c

OTHER OUTCOMES:
hypoglycemia (patient self report) | for the entire 6 month after start of the trial
  patient self report
Change in gut permeability (quantification of specific sugars in urine) | 3-month after start of the trial
  measure by amount of mannitol and lactulose in urine
Change in gut permeability (quantification of specific sugars in urine) | 6-month after start of the trial
  measure by amount of mannitol and lactulose in urine

CONTACTS AND LOCATIONS:
Overall Officials: Carol Huang, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ho J, Nicolucci AC, Virtanen H, Schick A, Meddings J, Reimer RA, Huang C. Effect of Prebiotic on Microbiota, Intestinal Permeability, and Glycemic Control in Children With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4427-4440. doi: 10.1210/jc.2019-00481. PMID 31188437
- [Derived] Ho J, Reimer RA, Doulla M, Huang C. Effect of prebiotic intake on gut microbiota, intestinal permeability and glycemic control in children with type 1 diabetes: study protocol for a randomized controlled trial. Trials. 2016 Jul 26;17(1):347. doi: 10.1186/s13063-016-1486-y. PMID 27456494